CLINICAL TRIAL: NCT03965702
Title: Impact of a Real Time Clinical Decision Support System to Guide Fluid Administration on Microvascular Parameters in Patients Undergoing Major Abdominal and Orthopedic Surgery: A Randomized Controlled Trial
Brief Title: Impact of an Assisted Fluid Management System on Microvascular Parameters
Acronym: MicroSupport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: APHP191024
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2021-12

CONDITIONS: Monitoring
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All microvascular parameters will be analyzed at the end of the study by a blinded physicians (not linked to the study and not author of the future manuscript)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EV1000 monitoring (Active Comparator): This group of patients will receive fluid administration during surgery based on a manual GDFT protocol actually in place in the department using the EV1000 monitoring device (Edwards Life sciences, Irvine, USA)
  Interventions: Other: Manual application of the GDFT protocol (standard of care)
- EV1000 monitoring with the decision (AFM) (Experimental): This group of patients will receive fluid administration during surgery based on a novel clinical decision support system for GDFT guidance using the EV1000 monitoring device (Edwards Life sciences, Irvine, USA)
  Interventions: Device: Use of a decision support system on the EV1000 monitoring (AFM mode)

INTERVENTIONS:
Device: Use of a decision support system on the EV1000 monitoring (AFM mode) — The way to administer fluid is based on the same monitoring device but will differ by the way fluid is given ( following a manual GDFT protocol versus following recommendation from an active clinical decision support system for fluid administration called AFM (assisted fluid management) Measurement of all microvascumlar parameters in blinded way. Blood pressure wil standardized in both group.
  Arms: EV1000 monitoring with the decision (AFM)
Other: Manual application of the GDFT protocol (standard of care) — Manual application of a GDFT protocol to guide fluid administration. Measurement of all microvascumlar parameters in blinded way. Blood pressure wil standardized in both group.
  Arms: EV1000 monitoring

SUMMARY:
This study will compare a group of patients managed with a manual GDFT protocol (using the EV1000 monitoring device; Edwards Life sciences, Irvine, USA) to a group of patients managed using a novel real time clinical decision support system for goal directed fluid therapy (GDFT) guidance on microvascular parameters in patients undergoing major abdominal or orthopedic surgery.

DETAILED DESCRIPTION:
Many trials have indicated that GDFT strategies may benefit high-risk surgical patients but these strategies are infrequently implemented on a day to day basis. It has also been shown that without any goal or protocol for fluid resuscitation, large inter- and intra-provider variability exist and have been correlated with marked variations in patient outcomes. Even under ideal study conditions, strict adherence to GDFT protocols is hampered by the workload and concentration required for consistent implementation.Haemodynamic monitors and protocols alone do not enable optimal fluid titration to be provided consistently to all patients - there must also be appropriate and timely interpretation and intervention.

To address this problem of consistency and protocol adherence, a novel real time clinical decision support system, "Assisted Fluid Management" (AFM), has been designed to help ease some of the workload associated with GDFT protocol implementation. The AFM system (released on the European market in March 2017) may help increase GDFT protocol adherence while leaving direction and guidance in the hands of the care providers. This system can suggest fluid bolus administration, analyse the effects of the bolus, and continually re-assess the patient for further fluid requirements.

Mean arterial pressure will be at least maintained in both groups above 65 mmHg with norepinephrine administration. Vasopressors administration is standardised in both groups (objective is a MAP of > 65 mmHg) and the only difference will be the way fluid boluses are given to the patient (following standard of care (manual protocol) of following the assisted fluid management recommandations)

A recent published study demonstrated that the implementation of the AFM for GDFT guidance resulted in a significantly longer period during surgery in a preload independent state (defined as a SVV < 13%) with a reduced total amount of fluid administered without any difference in postoperative complications.

Another recent study demonstrated that during abdominal surgery, microvascular perfusion is impaired during preload dependence (SVV >13%) and recovers after fluid administration (preload independent state)

Therefore the goal of this bicentric randomized controlled trial is to compare a manual GDFT approach (standard of care actually in the department) versus an Assisted fluid management approach (using the AFM mode) on the Microvascular flow index.

We assume that this novel clinical decision support system will allow patients to have less alterations of their microvascular parameters than patients managed under standard of care (GDFT but without the assisted fluid management mode)

ELIGIBILITY:
Inclusion Criteria:

* All adult patients in the operating room scheduled for a major abdominal & orthopedic surgery requiring a cardiac output monitoring (EV1000).
* Written informed consent received before surgery.

Exclusion Criteria:

* Minor Patients.
* No french speaking.
* Atrial fibrillation or severe arrythmia.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Microvascular flow index | Day 0
  Comparison of this index between groups during the intraoperative period. The image is divided into four quadrants and the predominant type of flow in very small vessels is assessed in each quadrant using an ordinal score (0= no flow; 1 = intermittent flow; 2 = sluggish flow; 3 = normal flow). The overall score, called microvascular flow index, is the sum of each quadrant score divided by the number of quadrants

SECONDARY OUTCOMES:
Composite criteria of minor postoperative complications | 30 days postsurgery
  This composite score includes 8 items (1 point for each item present; minimum score is 0 and maximum is 8 points)
  1. postoperative nausea and vomiting
  2. delirium and confusion
  3. Infection of surgical site
  4. urinary infection
  5. acute kidney injury (KDIGO I & II classiciation)
  6. paralytic ileus
  7. other infection (skin, catheter, unknown etc)
  8. Readmission to the hospital within 30 days postoperative
Composite criteria of major postoperative complications | 30 days postsurgery
  This composite score includes 14 items (one point for each item present; minimum score is 0 and maximum is 14 points):
  1. stoma dehiscence
  2. Peritonitis
  3. Sepsis
  4. wound dehiscence
  5. bleeding requiring a redo surgery
  6. pulmonary embolism
  7. pulmonary edema
  8. Pneumonia
  9. acute coronary syndrome
  10. atrial fibrillation
  11. stroke
  12. Dialysis
  13. non scheduled redo surgery
  14. 30days mortality (all causes)
Stroke volume over the procedure | Postoperative day 1
  average stroke volume over the procedure
Cardiac output over the procedure | Postoperative day 1
  average cardiac output over the surgery
Total Fluid received during the procedure | Postoperative day 1
  amount of fluid received during surgery
Net fluid balance | Postoperative day 1
  Net fluid balance at the end of the surgery
Hospital length of stay | 30 days postsurgery
  hospital length of stay
Proportion of perfused vessels | Day 0
  Comparison of this index between groups during the intraoperative period. This is calculated as follow: 100 x (total number of vessels - [no flow+intermittent flow]/total number of vessels.
Perfused vessel density | Day 0
  Comparison of this index between groups during the intraoperative period. This is calculated automatically by dividing the area of perfused vessels by the total area of interest using the Automated Vascular Analysis software.
Heterogeneity index | Day 0
  Comparison of this index between groups during the intraoperative period. This is calculated as follows: (highest site microvascular flow index-lowest site microvascular flow index) divided by the mean of the microvascular flow index of all sublingual sites.
minimal value of microvascular flow index | Day 0
  minimal value of this index during the intraoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, MD PhD, Principal Investigator — BICETRE HOSPITAL, APHP
Locations (1):
- Hôpital du Kremlin Bicêtre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coeckelenbergh S, Entzeroth M, Van der Linden P, Flick M, Soucy-Proulx M, Alexander B, Rinehart J, Grogan T, Cannesson M, Vincent JL, Vicaut E, Duranteau J, Joosten A. Assisted Fluid Management and Sublingual Microvascular Flow During High-Risk Abdominal Surgery: A Randomized Controlled Trial. Anesth Analg. 2025 May 1;140(5):1149-1158. doi: 10.1213/ANE.0000000000007097. PMID 39116013